CLINICAL TRIAL: NCT05385549
Title: A Phase 2 Study of 5 Years of Adjuvant Imatinib in Patients With Gastrointestinal Stromal Tumor With a High Risk of Recurrence Following Surgical Resection
Brief Title: 5 Years of Adjuvant Imatinib in Patients With Gastrointestinal Stromal Tumor With a High Risk
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC2202
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5 years of adjuvant imatinib treatment (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — Imatinib Mesylate, 400 mg once daily, oral. 5 years of adjuvant imatinib treatment (standard treatment 3years + IP treatment : 2yesrs)

SUMMARY:
In this study, the investigators aim to investigate the efficacy and safety of 5 years of adjuvant imatinib treatment in patients with tumor rupture defined by Nishida classification or those with a tumor size 10cm or larger and a mitotic index of 10/50HPFs or higher.

DETAILED DESCRIPTION:
Localized resectable GISTs can be cured with surgical resection, but no effective therapy had been established for patients with unresectable and/or metastatic GISTs and their prognosis was extremely poor before the advent of imatinib.

Imatinib mesylate is an oral tyrosine-kinase inhibitor (TKI) with activity against KIT, PDGFRA, ABL, and DDR. The efficacy of imatinib was first shown in the pivotal B2222 trial and confirmed by two subsequent randomized phase III trials. The standard dose of imatinib was established as a 400mg once daily dose upfront high-dose imatinib treatment with a 800mg daily dose showed a higher efficacy in terms of progression-free survival (PFS) in patients with GISTs harboring KIT exon 9 mutations but also higher toxicity. The median time-to-progression (TTP) with imatinib was about 2 years in the extended follow-up results of the B2222 trial. Imatinib efficacy correlates with primary KIT mutations and patients with KIT exon 9 mutations had worse survival outcomes than those with KIT exon 11 mutations.

Surgical resection is the mainstay of the treatment of localized GIST. However, in a proportion of patients, a high recurrence rate was observed, which prompted the investigation of the clinical efficacy of adjuvant imatinib treatment. The ACOSSOG Z9001 study showed that one year of adjuvant imatinib treatment after surgical resection in patients with a tumor size of 3cm of larger improved recurrence-free survival compared to placebo. This study was the first to demonstrate the efficacy of adjuvant imatinib treatment. Subsequently, SSG XVIII/AIO study showed that 3 years of adjuvant imatinib improved recurrence-free survival and overall survival compared to one year of adjuvant imatinib in High risk patients defined by modified NIH criteria. Based on this study in patients classified as high risk by the modified NIH criteria, 3 years adjuvant imatinib is the standard of care.

However, given that a substantial proportion of such patients show disease recurrence, the PERSIST5 study recently showed that 5 years of imatinib treatment may further reduce the recurrence. In addition, clinical outcomes of the patients classified as high risk by the modified NIH criteria are heterogeneous, and some of these patients show particularly poor clinical outcomes. The investigators analyzed the clinical outcomes of 222 high risk GIST patients who received 3 years of adjuvant imatinib treatment following surgical resection. Among these, patients with tumor rupture defined by Nishida classification or those with a tumor size 10cm or larger and a mitotic index of 10/50HPFs or higher had poor clinical outcomes with a 5-year recurrence-free survival of 50%.

In this study, the investigators aim to investigate the efficacy and safety of 5 years of adjuvant imatinib treatment in patients with tumor rupture defined by Nishida classification or those with a tumor size 10cm or larger and a mitotic index of 10/50HPFs or higher.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or older, at the time of acquisition of informed consent
2. Histologically confirmed GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
3. (1) Completely resected localized GIST (R0 resection) within 12 weeks prior to the start of the adjuvant imatinib.

(2) After complete resection(R0 resection), High risk GIST according to Modified NIH criteria and ongoing adjuvant imatinib treatment.

4) High risk GIST according to Modified NIH criteria,

1. Tumor rupture according to Nishida classification or
2. tumor size >10cm and mitosis >10/50 HPF 5) Eastern Cooperative Oncology Group (ECOG) performance status 0 ~ 2 6) Adequate bone marrow, hepatic, renal, and other organ functions, before adjuvant imatinib treatment

   * Neutrophil >1,500/mm3
   * Platelet > 100,000/mm3
   * Hemoglobin >8.0 g/dL
   * Total bilirubin < 1.5 x upper limit of normal (ULN)
   * AST/ALT < 2.5 x ULN
   * Creatinine <1.5 x ULN 7) Provision of a signed written informed consent

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breast feeding
2. Women or men who are not willing to use effective contraception entering the study period or until at least 3 months after the last study drug administration.
3. If any of the following applies within ≤ 6 months prior to starting study enrollment : Myocardial Infarction, severe instable angina, coronary/peripheral bypass, NYHA class III or IV congestive heart failure, stroke or transient ischemic attack, treatment required severe arrhythmia.
4. Uncontrolled infection
5. Acute and chronic liver disease and all chronic liver impairment.(But Patients with stable chronic hepatitis B are eligible)
6. Patients who had reduced the dose of imatinib to less than 300 mg/day due to toxicity.
7. Acute, or chronic medical or psychiatric condition or laboratory abnormality such as active uncontrolled infection that difficult to study participation in the judgment of the investigator
8. Known diagnosis of HIV infection (HIV testing is not mandatory).
9. History of another primary malignancy that is currently clinically significant or currently requires active intervention.
10. Alcohol or substance abuse disorder.
11. The patients with PDGFRα D842V mutation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 5years
  Progression-free survival (PFS) per the RECIST v1.1 is defined as the time from the date of first dosing of Imatinib to the date of progression or death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Seoul, South Korea